CLINICAL TRIAL: NCT02411682
Title: Effect of Breakfast on Overall Postprandial Hyperglycemia in T2D
Brief Title: Breakfast on Postprandial Hyperglycemia
Acronym: B-PPHG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas Caracas (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Daniela Jakubowicz, MD, Prof. Daniela Jakubowicz MD, Hospital de Clinicas Caracas
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: HCCBI 057-2013-254
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- YesB (Active Comparator): On YesB day the patients will consume breakfast , lunch and dinner
  Interventions: Other: Breakfast eating (YesB); Other: Breakfast skipping (NoB)
- NoB (Experimental): On NoB Day The patient will consume only lunch and dinner
  Interventions: Other: Breakfast eating (YesB); Other: Breakfast skipping (NoB)

INTERVENTIONS:
Other: Breakfast eating (YesB) — On YesB day the patients will eat Breakfast at 8:00, Lunch at 13:30 and Dinner at 19:00
Other: Breakfast skipping (NoB) — On NoB day the patients will fast until lunch, then will eat Lunch at 13:30 and Dinner at 19:00

SUMMARY:
Reduction of postprandial hyperglycemia (PPHG) is a major target in the treatment of type 2 diabetes (T2D). Skipping breakfast has been consistently associated with higher HbA1c and overall PPHG in subjects with type 2 diabetes (T2D). Our aim was to explore the effect of skipping vs eating breakfast on PPHG after subsequent isocaloric (700kcal) lunch and dinner

DETAILED DESCRIPTION:
In type 2 diabetic individuals the omission of breakfast is associated with significant increase in HbA1C and all-day postprandial hyperglycemia even without overeating in the evening. In contrast, high-energy breakfast and low-energy dinner result in a significant reduction of all-day postprandial glycaemia Similarly, 3 months of high-energy breakfast led to a 5% reduction in HbA1C levels in type 2 diabetes participants Despite the growing evidence showing the beneficial effects of breakfast consumption on overall postprandial hyperglycemia and HbA1C levels, very little is known regarding the relationship between breakfast skipping and all-day glycemic excursions in type 2 diabetes patients. Therefore, to test whether breakfast skipping influences metabolic responses to the following meals in type 2 diabetes patients during the same day, we explored the postprandial glycemic response to identical lunch and dinner meal tests with or without breakfast.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 26-34 kg/m2.
* HbA1c > 7 %
* T2D since < 10 yrs,
* . Only non treated or treated with oral antidiabetic drugs
* Those treated with insulin or GLP-1 analogs will be excluded.

Exclusion Criteria:

* Type 1 diabetes
* Serum creatinine level > 1.5 mg/dl
* Pulmonary disease, psychiatric, immunological, neoplastic diseases or severe diabetic complications,such as cardiovascular disease, cerebrovascular disease, proliferative diabetic retinopathy, gastroparesis or anemia (Hg > 10g/dL) or underwent bariatric surgery.
* Abnormal liver function tests
* Participating in dietary program or using of weight-loss medications
* History (within one year) of illicit drug abuse or alcoholism.
* Use of psychotropic or anoretic medication during the month immediately prior to study onset

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Postprandial Glucose | 6 weeks
  Postprandial Glucose will be measure after lunch and dinner

SECONDARY OUTCOMES:
Postprandial intact GLP-1 | 6 weeks
  Postprandial intact GLP-1 will be measure after lunch and dinner
Postprandial Insulin | 6 weeks
  Postprandial Insulin will be measure after lunch and dinner
Postprandial Glucagon | 6 weeks
  Postprandial Glucagon will be measure after lunch and dinner
Postprandial Free Fatty Acids | 6 weeks
  Postprandial Free Fatty Acids will be measure after lunch and dinner

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Jakubowicz, MD, Principal Investigator — Hospital de Clinicas Caracas; Daniela Jakubowicz, MD, Principal Investigator — E. Wolfson Medical Center. Israel